CLINICAL TRIAL: NCT00189332
Title: Pilot Phase II, Open Label, Multicenter, Efficacy and Safety Study of 852A Administered Intravenously to Subjects With Unresectable Metastatic Cutaneous Melanoma.
Brief Title: Use of 852A in Metastatic Cutaneous Melanoma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1527-852A
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2008-10-27 (Estimated); Status verified 2008-10

CONDITIONS: Melanoma; Unresectable Metatstatic Cutaneous Melanoma
Keywords: Oncology; Melanoma
MeSH Terms: conditions — Melanoma; Neoplasms

INTERVENTIONS:
Drug: 852A

SUMMARY:
Pilot study to test the efficacy of 852A administered intravenously up to 3 times per week for 12 weeks in subjects with inoperable metastatic cutaneous melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Advanced melanoma not responding to 1st line chemotherapy
* Histological evidence of melanoma
* Measurable disease according to RECIST criteria
* ECOG performance status less than or equal to 2
* Life expectancy 6 months or more
* Normal organ and bone marrow function as defined by hematological and serum chemistry limits
* Adequate contraception for females of childbearing potential

Exclusion Criteria:

* Stage IV disease which has previously progressed during interferon treatment.
* Restriction of some therapies/medications for a certain timeframe prior to enrollment and during the study including: investigational drugs, high dose corticosteroids, immunotherapy, immunosuppressive medications, radiotherapy and drugs known to prolong QT interval and/or induce Torsades De Pointes
* History of uncontrolled seizure disorders
* Uncontrolled coagulation disorders.
* History or evidence of myocardial ischemia, congestive heart failure or arrythmias requiring treatment in the past 6 months
* History of uncontrolled intercurrent or chronic illness
* Concurrent malignancies.
* Brain metastases.
* HIV positive.
* Prolonged QTc interval
* Uncontrolled intercurrent or chronic illnesses.
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2005-02; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
assessing antitumor activity of 852A intravenous bolus injection administered 3 times a week for 12 weeks

SECONDARY OUTCOMES:
to assess the safety of the dosage regiment over 12 weeks
to obtain preliminary data regarding the safety and long term efficacy of 852A in subjects treated with the drug for more than 12 weeks

CONTACTS AND LOCATIONS:
Locations (8):
- France (2):
  - Hôpital Hotel Dieu, 1, Pace de l' Hôpital,, Lyon
  - Hôpital Ste Marguerite,Service de Dermatologie, Marseille
- Germany (5):
  - Hautklinik, Medizinische Einrichtungen der Heinrich-Heine - Universität Düsseldorf, Düsseldorf
  - Klinik und Poliklinik für Dermatologie und Venerologie Universitätsklinikum Essen, Essen
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - (DKFZ) an der Universitäts-Hautklinik Mannheim, Mannheim
  - Universitätsklinik und Poliklinik für Hautkrankheiten, Würzburg
- Universitatsspital Zurich, Zurich, Switzerland